CLINICAL TRIAL: NCT02186353
Title: Effect of Intact vs. Highly Processed Whole Grains on Insulin Sensitivity and Other Cardiometabolic Risk Factors in Hyperinsulinemic Adults
Brief Title: Processing Responses of Grains (PRO-Grains) Study
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of adequate funding
Sponsor: Boston Children's Hospital (Other)
Collaborators: Kansas State University (Other)
Responsible Party: Principal Investigator, Julia Wong, Instructor in Pediatrics, Boston Children's Hospital
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: P00009343
Record Dates: First submitted 2014-06-17; First posted 2014-07-10 (Estimated); Last update posted 2017-04-11 (Actual); Status verified 2017-04

CONDITIONS: Insulin Resistance; Cardiovascular Disease; Diabetes
Keywords: Whole grains; Food processing; Cardiometabolic risk factors
MeSH Terms: conditions — Insulin Resistance; Cardiovascular Diseases; Diabetes Mellitus

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (3):
- Intact/minimally processed whole grains (Experimental): Partial feeding study
  Interventions: Behavioral: Partial feeding study
- Highly processed whole grains (Experimental): Partial feeding study
  Interventions: Behavioral: Partial feeding study
- Refined grains (Active Comparator): Partial feeding study
  Interventions: Behavioral: Partial feeding study

INTERVENTIONS:
Behavioral: Partial feeding study — Provision of all grain foods where only the processing of kernels used to produce the grain foods will differ among test diets. Each participant will be assigned to complete the three 4-week test diets in random sequence.

SUMMARY:
The primary objective of this pilot study will be to examine the effects of consuming whole grains, differing in the degree of processing, on insulin sensitivity and other cardiometabolic risk factors. The overall aim will be to assess feasibility of the test diets and to generate preliminary data.

DETAILED DESCRIPTION:
In this pilot study, the investigators will access feasibility and generate preliminary data to systematically address a major question in nutrition: Does food processing, specifically with regard to whole grains (WGs), have an independent effect on outcomes related to diabetes and cardiovascular disease? Whole grains are defined as intact, ground, cracked, or flaked caryopsis (kernel or seed), where the principal components (bran, endosperm, germ) are present in the same proportion as the intact caryopsis. In contrast, refined grains (RGs) are milled to remove the bran and germ, leaving only the endosperm and resulting in lower fiber, iron, and many B vitamins. Several previous studies have shown that consumption of WGs vs. RGs improves insulin sensitivity and decreases risk for chronic disease. However, the effects of consuming WGs may differ depending on degree of processing. While whole grain products contain the three components of the kernel, we hypothesize that consuming the food containing the least processed (and least pulverized) kernels may have beneficial effects on metabolism that decrease disease risk through plausible physiological mechanisms.

The investigators propose a partial feeding study using a randomized 3-period crossover design to compare the effects of 1) intact or minimally processed whole grains, 2) highly processed whole grains, and 3) refined grains, each fed for 4 weeks. The primary outcome will be change in peripheral insulin sensitivity. Secondary outcomes include hepatic insulin sensitivity, components of the metabolic syndrome and other cardiometabolic risk factors, arterial stiffness, gut microbiome and fecal short chain fatty acids, and ratings of hunger, satiation, palatability, and acceptability (gastrointestinal symptoms).

ELIGIBILITY:
Inclusion Criteria:

* Aged 18 to 35 years
* Body mass index ≥ 25 and <40 kg/m2
* Serum fasting insulin >10 uIU/mL and one of the following metabolic syndrome components: waist circumference, men: ≥102 cm, women: ≥88 cm; triglycerides, ≥150 mg/dL; HDL-C, men: <40 mg/dL , women: <50 mg/dL; systolic blood pressure ≥130 or diastolic blood pressure ≥85 mmHg; or fasting glucose, ≥100 mg/dL
* Medical clearance from a primary care provider to rule out any major medical illness, disability, or disorder (e.g., liver disease, renal failure, cancer)
* Access to a working telephone or cell phone
* Willingness to eat the grain foods provided during participation
* If female, regular menstrual cycles (defined as 26-30 days, ±1 day full flow, i.e. 26 to 30 days between cycles; no more than one day variation in the duration of menstrual flow)

Exclusion Criteria:

* Pre-existing major medical illness by medical history or laboratory screening tests
* Allergy or sensitivity to gluten (self-reported or physician diagnosed)
* >5% change in weight within previous 6 months
* Current smoking (1 cigarette in the past week)
* Major surgery within the previous 6 months
* Physical, mental, or cognitive handicaps that prevent participation.
* Alcohol intake >7 drinks per week
* Use of medications that may affect study outcomes
* Use of antibiotics within the previous 3 months (in those who agree to complete the analyses of gut microbiome and fecal short chain fatty acids)
* Use of illegal drugs
* Plans to be away from home for 1 week or longer during the study period (e.g., vacation, relocation)
* Another member of the family (first degree relative) or household participating in the study
* If female, pregnancy or lactation during prior 12 months, plans to become pregnant during the study period, change in oral contraceptives within 3 months, or irregular menstrual cycle frequency (<10 bleeds/year)

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2014-09; Primary Completion 2015-09 (Estimated); Study Completion 2015-09 (Estimated)

PRIMARY OUTCOMES:
Change from week 0 in peripheral insulin sensitivity (assessed by frequently-sampled oral glucose tolerance test) at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in peripheral insulin sensitivity (assessed by frequently-sampled oral glucose tolerance test) at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in peripheral insulin sensitivity (assessed by frequently-sampled oral glucose tolerance test) at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)

SECONDARY OUTCOMES:
Change from week 0 in hepatic insulin sensitivity (assessed by frequently-sampled oral glucose tolerance test) at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in hepatic insulin sensitivity (assessed by frequently-sampled oral glucose tolerance test) at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in hepatic insulin sensitivity (assessed by frequently-sampled oral glucose tolerance test) at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in fasting glucose at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in fasting glucose at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in fasting glucose at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in fasting insulin at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in fasting insulin at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in fasting insulin at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in blood lipids at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in blood lipids at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in blood lipids at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in high-sensitivity C-reactive protein at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in high-sensitivity C-reactive protein at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in high-sensitivity C-reactive protein at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in plasminogen activator inhibitor-1 (PAI-1) at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in plasminogen activator inhibitor-1 (PAI-1) at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in plasminogen activator inhibitor-1 (PAI-1) at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in alanine aminotransferase (ALT) at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in alanine aminotransferase (ALT) at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in alanine aminotransferase (ALT) at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in serum metabolomics profile at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in serum metabolomics profile at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in serum metabolomics profile at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in blood pressure at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in blood pressure at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in blood pressure at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in waist circumference at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in waist circumference at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in waist circumference at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in arterial stiffness (assessed by carotid-femoral pulse wave velocity) at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in arterial stiffness (assessed by carotid-femoral pulse wave velocity) at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in arterial stiffness (assessed by carotid-femoral pulse wave velocity) at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in gut microbiome composition (16s rRNA sequencing) and fecal short chain fatty acids at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in gut microbiome composition (16s rRNA sequencing) and fecal short chain fatty acids at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in gut microbiome composition (16s rRNA sequencing) and fecal short chain fatty acids at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in ratings of hunger and satiation at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in ratings of hunger and satiation at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in ratings of hunger and satiation at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in ratings of palatability and acceptability (gastrointestinal symptoms) at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in ratings of palatability and acceptability (gastrointestinal symptoms) at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in ratings of palatability and acceptability (gastrointestinal symptoms) at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in body weight at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in body weight at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in body weight at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in dietary intake at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in dietary intake at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in dietary intake at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in physical activity (assessed by accelerometry) at week 4 | Week 0, Week 4 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in physical activity (assessed by accelerometry) at week 8 | Week 0, Week 8 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)
Change from week 0 in physical activity (assessed by accelerometry) at week 12 | Week 0, Week 12 (End of 4-week diet of intact/minimally processed whole grains OR highly processed whole grains OR refined grains)

CONTACTS AND LOCATIONS:
Overall Officials: Julia MW Wong, PhD, RD, Principal Investigator — Boston Children's Hospital; David S Ludwig, MD, PhD, Study Chair — Boston Children's Hospital; Cara B Ebbeling, PhD, Study Chair — Boston Children's Hospital
Locations (1):
- Children's Hospital Boston, Boston, Massachusetts, United States